CLINICAL TRIAL: NCT05569824
Title: Evaluating the Test Performance of Aspergillus Antigen Detection Using a Lateral-flow Device (LFD) on Broncho-alveolar Lavage (BAL) Fluid for the Diagnosis of Invasive Pulmonary Aspergillosis in Paediatrics: A Pilot Study
Brief Title: LFD of Aspergillus Antigen in Paediatrics
Acronym: LFD-AsPaeds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); University College, London (Other); St George's, University of London (Other); Fungal Infection Trust (Unknown)
Responsible Party: Sponsor
Organization: St George's, University of London (Other)
Other Study IDs: 292170
Record Dates: First submitted 2022-08-17; First posted 2022-10-06 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Invasive Pulmonary Aspergillosis; Invasive Fungal Disease
Keywords: Lateral-flow Device; Aspergillus; Broncho-alveolar Lavage; Invasive Pulmonary Aspergillus; Paediatrics; Aspergillus Antigen Detection; Invasive Fungal Disease
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Bronco-alveolar lavage (BAL) fluid will be collected.
  If participants/parents/legal guardians provide consent
  Participants/parents/legal guardians can provide consent to the
  the anonymised samples will be stored for future ethically approved research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Study Pathway: Child or young person undergoing a Broncho-alveolar Lavage (BAL) for suspected pulmonary Invasive Fungal Disease (IFD) and consent obtained.
  Interventions: Diagnostic Test: Lateral-flow Device

INTERVENTIONS:
Diagnostic Test: Lateral-flow Device — An additional amount of 0.1-0.2 ml (2-4 drops) of bronco-alveolar lavage (BAL) fluid will be collected during the bronchoscopy which is carried out as part of the standard of care. The LFD test will be carried out on the BAL fluid collected.

SUMMARY:
Many children and young people are at risk of invasive fungal disease (IFD), such as those who have had a haematopoietic stem cell transplants, those with an immune deficiency or those who are prescribed immunosuppressive drugs, for example, corticosteroids. One type of mould that causes invasive fungal disease is called Aspergillus. There is currently no quick test which can tell us if someone has an invasive fungal disease caused by Aspergillus called Aspergillosis. It is a difficult condition to diagnose and the results from the tests that are involved take days or weeks to come back. These tests including a few different blood tests, a scan of the lungs (CT scans) and taking fluid from inside the lungs/airway.

A new test for Aspergillosis is the lateral flow device (LFD) assay. This is a rapid test which gives a result within minutes. It involves testing a sample of the fluid from the lungs/airway. This fluid can be obtained as part of the routine investigations for Aspergillosis. It has been shown to be a good and safe test in adults but the investigators do not know if it will be a valuable test in children and young people yet. The purpose of this study is to determine whether the LFD test can effectively diagnose Aspergillosis in children and young people.

DETAILED DESCRIPTION:
The overall study design is a prospective, single centre, cohort study in patients who have suspected pulmonary Invasive Aspergillosis (IA)/IFD and hence have a diagnostic BAL as part of their clinical care. A total number of 20 children <18 years of age undergoing a BAL for suspected IA/IFD at St George's Hospital University Hospitals NHS Foundation Trust (United Kingdom) will be enrolled. No changes in the regular diagnostic pathway or treatment will be done for this study.

If patients are scheduled to have a BAL sample and meet the Inclusion/Exclusion criteria the patients will be approached for consent at the same time as consent for the standard of care BAL procedure. With the patients consent the samples will be retrieved from the BAL fluid, both for the standard of care investigations (fungal culture, GM and fungal PCR in BAL fluid) and for the study sample. The minimal study sample required will be 1 ml. The study samples will be tested directly with the LFD for Aspergillus antigen when possible. Haemorrhagic or too viscous samples will need to be previously treated with a buffer (150 ul BAL with 300 ul buffer). Every individual participant patient will be followed up prospectively at two weeks and 3-months post-BAL to collate information.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients aged less than 18 years who are clinically identified as requiring investigation for pulmonary IA/IFD and hence are undergoing a BAL as part of clinical care
* Written informed consent

Exclusion Criteria:

* Patients who are undergoing a BAL for other indications than suspected invasive fungal lung disease
* Patients ≥ 18 years of age

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients undergoing a BAL for suspected IA/IFD at St George's University Hospitals NHS Foundation Trust (United Kingdom).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-01-19 (Estimated); Study Completion 2024-04-29 (Estimated)

PRIMARY OUTCOMES:
The proportion of children whose diagnosis has been supported by the LFD test | Through study completion, an average of 2 years
The sensitivity of test results compared to culture and PCR results | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ferreras-Antolin, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (1):
- St George's University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.